CLINICAL TRIAL: NCT06930391
Title: Effect of Extracellular Calcium on Carbetocin Mediated Contractility in Human Myometrium: An Ex-Vivo Study
Brief Title: Effect of Extracellular Calcium on Carbetocin Mediated Contractility in Human Myometrium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-01
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Hemorrhage (Primary)
Keywords: carbetocin; calcium; uterine contraction; cesarean delivery
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carbetocin; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Calcium 1.25nM with NO oxytocin pre-exposure (Active Comparator): Dose-response testing with 1.25nM calcium chloride, and increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-10 M to 10-5 M, with NO oxytocin pre-exposure
  Interventions: Drug: Carbetocin; Drug: Calcium
- Calcium 2.5nM with NO oxytocin pre-exposure (Active Comparator): Dose-response testing with 2.5nM calcium chloride, and increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-10 M to 10-5 M, with NO oxytocin pre-exposure
  Interventions: Drug: Carbetocin; Drug: Calcium
- Calcium 5.0nM with NO oxytocin pre-exposure (Active Comparator): Dose-response testing with 5.0nM calcium chloride, and increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-10 M to 10-5 M, with NO oxytocin pre-exposure
  Interventions: Drug: Carbetocin; Drug: Calcium
- Calcium 1.25nM with oxytocin pre-exposure (Active Comparator): Dose-response testing with 1.25nM calcium chloride, and increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-10 M to 10-5 M, with oxytocin pre-exposure
  Interventions: Drug: Oxytocin; Drug: Carbetocin; Drug: Calcium
- Calcium 2.5nM with oxytocin pre-exposure (Active Comparator): Dose-response testing with 2.5nM calcium chloride, and increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-10 M to 10-5 M, with oxytocin pre-exposure
  Interventions: Drug: Oxytocin; Drug: Carbetocin; Drug: Calcium
- Calcium 5.0nM with oxytocin pre-exposure (Active Comparator): Dose-response testing with 5.0nM calcium chloride, and increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-10 M to 10-5 M, with oxytocin pre-exposure
  Interventions: Drug: Oxytocin; Drug: Carbetocin; Drug: Calcium

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 10-5M will be added to 3 groups of myometrial strips for 2 hours to induce desensitization.
  Arms: Calcium 1.25nM with oxytocin pre-exposure; Calcium 2.5nM with oxytocin pre-exposure; Calcium 5.0nM with oxytocin pre-exposure
Drug: Carbetocin — Increasing concentrations of carbetocin in a pattern of 1 log molar increase every 10 min, from 10-10 M to 10-5 M
Drug: Calcium — Calcium chloride in the following concentrations:1.25mM, 2.5mM and 5.0mM.

SUMMARY:
Postpartum hemorrhage (PPH) continues to be an increasing problem globally. Uterotonics play an essential role in the pharmacological management of uterine atony. Carbetocin, a long acting analog of oxytocin has been recommended as a first line uterotonic for PPH prophylaxis at cesarean delivery. Considering many woman have associated comorbidities and are at high risk of PPH, finding alternative pharmacological agents is essential. Calcium is a key factor for myometrial contractions and calcium blood levels can be low at the end of pregnancy. Both hypocalcemia and hypercalcemia could lead to a decrease in myometrial contractions. It is already been demonstrated that in both desensitized and naïve myometrium, normocalcemia provides a better uterine tone compared to hypo and hypercalcemia when oxytocin is given as the first uterotonic drug.

Currently, the role of extracelullar calcium in carbetocin- induced contractility is unknown. This will be the first ex vivo study to test the effects of extracellular calcium on oxytocin pretreated and naive myometrium. The results of this study will provide evidence on the use of this safe drug in clinical practice, particularly in women with labour arrest, and provide alternative pharmacological strategies to both prevention and treatment of PPH, thus improving our clinical practice.

The investigators hypothesize that extracellular normocalcemia would provide superior carbetocin-mediated contractility in both naive and oxytocin-pretreated myometrium compared with hypercalcemia and hypocalcemia.

ELIGIBILITY:
Inclusion Criteria:

* non-laboring women with gestational age between 37 to 41 weeks
* not exposed to exogenous oxytocin, scheduled for a primary or first repeat cesarean delivery under neuraxial anesthesia.

Exclusion criteria:

* patients requiring general anesthesia
* more than 1 previous cesarean delivery
* history of uterine atony
* emergency cesarean section in labor
* patients using medications that could affect myometrial contractility such as nifedipine, labetalol, or magnesium sulphate.
* patients with any condition of predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, severe preeclampsia, macrosomia, polyhydroamnios, large uterine fibroids, chorioamnionitis, previous history of postpartum bleeding.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Motility index | 4 hours
  Motility index (MI) is a calculated outcome, based on the formula: frequency/(10 x amplitude). Frequency and amplitude are secondary outcome measures as described below. The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 4 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 4 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist. The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No